CLINICAL TRIAL: NCT04583072
Title: SEPTA Trial: Stockholm3 Validation Study in a Multi-Ethnic Cohort for ProsTAte Cancer
Brief Title: Stockholm3 Validation Study in a Multi-Ethnic Cohort
Acronym: SEPTA
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: University of Illinois at Chicago (Other); UroPartners (Unknown); University of Chicago (Other); Rush University Medical Center (Other); Montefiore Medical Center (Other); The University of Texas Health Science Center at San Antonio (Other); Cook County Health & Hospitals System (Other); Cook County Health (Other Government); Stanford University (Other); Northwestern Medicine (Other); University of Southern California (Other); University Health Network, Toronto (Other); Urology Clinics of North Texas (Network); LAC+USC Medical Center (Other)
Responsible Party: Principal Investigator, Henrik Grönberg, Professor, Karolinska Institutet
Other Study IDs: KarolinskaI3
Record Dates: First submitted 2020-09-28; First posted 2020-10-12 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer (Diagnosis)
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venipuncture: Prior to the biopsy the blood will be collected in 2 EDTA (lavender top) x 4 milliliters (8 milliliters total) tubes will be removed after obtaining consent from the subjects. One tube will be immediately centrifuged (10 minutes at 2000G) and plasma decanted to a tube without additives (this typically produces approximately 1.5 milliliters of plasma). The decanted tube (with plasma) and the remaining EDTA tube (with whole blood) is then frozen and stored at -20 degrees Celsius until being shipped to the A3P lab for Stockholm3 testing and analysis at -20 degrees Celsius (unless processing for DNA extraction and plasma analysis).
  Other biobanked specimens (as described in the Study detailed description) will be collected prospectively and will include plasma and Buffy Coat (used for DNA extraction) utilising the study inclusion and exclusion criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-Hispanic/Latino White/Caucasian men: Self-identified as White Non-Hispanic men, with age range (45.0 - 75.0 years), without prior evidence of prostate cancer
  Interventions: Diagnostic Test: The Stockholm3 test
- African/Black men: Self-identified as African or Black men, with age range (45.0 - 75.0 years), without prior evidence of prostate cancer
  Interventions: Diagnostic Test: The Stockholm3 test
- Hispanic/Latino White/Caucasian men: Self-identified as White Hispanic men, with age range (45.0 - 75.0 years), without prior evidence of prostate cancer
  Interventions: Diagnostic Test: The Stockholm3 test
- Asian men: Self-identified as Asian men, with age range (45.0 - 75.0 years), without prior evidence of prostate cancer
  Interventions: Diagnostic Test: The Stockholm3 test

INTERVENTIONS:
Diagnostic Test: The Stockholm3 test — Venipuncture: Prior to the biopsy the blood will be collected in 2 EDTA (lavender top) x 4 ml tubes will be removed after obtaining consent from the subjects.
  Other Names: Diagnostic Test: Custom ancestry informative genetic markers

SUMMARY:
Introduction: Prostate cancer (PCa) is the most commonly detected cancer in men and is the second leading cause of cancer death. Differences in race and ethnicity have been shown to have differences in PCa incidence, detection, and outcomes. Current prostate cancer screening involves prostatic specific antigen (PSA) which is a nonspecific protein marker (aka kallikrein) that can often leads to unnecessary biopsies (up to 74% benign biopsies) and clinical overdiagnosis (with up to 22% clinically insignificant cancer). Recently more sophisticated tests have been developed for PCa screening in the United States such as the Prostate Health Index (PHI) and the 4k (kallikrein) score, as well as clinical models that use information from the patient clinical history. However, these tests utilize limited serum protein assays and none of the established screening protocols utilize genetic variables to help account for the likely inherited risks as seen in different ethnicities.

A recent Swedish, prospective, population-based study, published in the Lancet Oncology, developed a unique multivariable biopsy outcome prediction model within a Nordic population of nearly 60,000 men. This model, the Stockholm3, which incorporated plasma protein markers, germline DNA SNPs as well as clinical variables, was shown to be capable of reducing the number of biopsies by 44% compared to PSA while maintaining adequate sensitivity for detection of PCa.

It is unknown whether an approach developed in Sweden that incorporates protein markers, genetics, clinical variables, and genetic ancestry would be beneficial in a racially diverse cohort.

Hypothesis: The investigators hypothesize that, a prospectively studied multiethnic cohort of men with the Stockholm3 test will identify unique and common risk factors that improve prostate cancer detection.

Aim: To assess the performance of the Stockholm3 test as compared to PSA and to identify unique features associated with PCa in Black/African American (n=500), Asian (n=500), White/Caucasian Hispanic (n=500), and White/Caucasian Non-Hispanic (n=500) men.

Methods: The investigators propose a prospectively identified cohort with participating institutions which have screened positive to undergo a prostate biopsy to have a retrospective analysis the Stockholm3 test and ancestry markers. Within this cohort the investigators will examine several predetermined risk factors to investigate their relationship to prostate cancer.

This blood sample will be tested for quantitative levels of serum protein markers and DNA will be extracted and will be tested for germline mutations as defined by the Stockholm3 test and other ancestry informative markers. Results from the study will be presented in such a way that no individual information will be disclosed.

DETAILED DESCRIPTION:
Study Design and Procedures:

The research coordinator will explain the information contained within the consent. Additionally, patient's blood will be drawn prior to their biopsy.

Prior to the biopsy, blood will be collected in x2 ethylenediaminetetraacetic acid (EDTA) 4 ml tubes after obtaining consent from the subjects. One tube will be immediately centrifuged (10 minutes at 2000G) and plasma decanted to a tube without additives (this typically produces 1.5 ml of plasma). The decanted tube (with plasma) and the remaining EDTA tube (with whole blood) is then frozen and stored at the designated participating institutional site. It will be stored at -20 Celsius until being shipped. The SEPTA specific blood collection is followed by the following collaborators: Uropartners, University of Illinois at Chicago, University of Chicago, Rush Medical Center, Montefiore, University of Texas Health Science Center of San Antonio, Urology Clinics of North Texas, University of Southern California Keck School of Medicine, Los Angeles County Hospital, Stanford University.

Additional samples from University Health Network (Toronto), Northwestern Medicine, John H. Stroger, Jr. Hospital of Cook County, and Cook County Health System (Chicago) will be included from biobanked sources which were prospective collected meeting inclusion and exclusion criteria.

Patient data will be stored in a REDCap database, hosted on Sweden's secure server. Data will be stored for the duration of the study, and 5 years afterwards for data analysis purposes.

Consented patients will be tracked by patient logs by each participating institution. The medical record number will be collected to keep a consistent identifier for data collection by key site personnel. Once all the patient data is recorded the data will be exported from REDCap with the MRN removed. There will be no patient identifiers used at the Karolinska Institute or A3P lab. The following PHI and non-PHI information will be logged of the patient:

PHI:

Medical record number (MRN)

Non-PHI Demographic data

* Stockholm3 Identification number
* Race
* Zip code

Clinical data

* Total PSA
* Age on sampling date [years]
* Family history of prostate cancer
* Use of 5-alpha reductase inhibitors
* Earlier biopsy conducted
* Prostate volume [Prostate volume as measure with US]
* Digital rectal exam status [Benign/normal, Nodule/induration felt, Asymmetry, Not performed]

AND

Outcome data - Results from biopsy performed immediately after blood venipuncture, i.e.:

Results will be separated into targeted biopsy cores and systematic biopsy cores

* Gleason Score 1
* Gleason Score 2
* Gleason Sum
* Cancer length (mm) (total and highest grade)
* Number of cores
* Number of positive cores
* Time to perform biopsy after blood draw [days]
* Results from MRI, i.e. Prostate Imaging Reporting & Data System (PIRADS) (0, 1, 2, 3, 4, 5)

Permitted use:

To run the Stockholm3 test defined by Gronberg et al AND Ancestry informative genetic markers

Samples will be shipped to the Uppsala based laboratory (A23 Laboratory) in Sweden for analysis. Each patient will have two blood samples (plasma and whole blood) and will be frozen at -20 Celsius. The blood samples will then be tested for quantitative levels of serum protein levels and DNA will be extracted from white blood cells and will be tested for gene and small nucleotide polymorphic (SNPs) germline mutations and variants .

Genotyping will be performed using custom genotyping assays. Plasma will be used for protein analysis. Plasma protein analysis will be performed using a custom protein assays including total and free PSA, human glandular kallikrein 2 (hK2), microseminoprotein-beta (MSMB), and Macrophage inhibitory cytokine 1 (MIC-1). PSA will be tested with a commercial assay.

Based on the results from the plasma protein analysis, the genetic analysis and clinical data, the Stockholm3 Risk Score will be calculated. The participants' samples will be treated in accordance with the regulations of Sweden at the laboratory based in Uppsala, Sweden.

Results of the tests will not be shared with the patient, nor will the results change or impact medical decisions.

Expected Risks/Benefits

Anticipated Risks:

As this is retrospective analysis of deidentified patient information as well as deidentified biospecimens, there are few anticipated risks. A confidentiality breach as well as loss of privacy are possible, however every effort will be made to minimize this risk.

Anticipated Benefits:

Participants will advance scientific and clinical knowledge. Participants will also receive a small payment for the time and involvement in the study.

Data Collection and Management Procedures

This study will utilize REDCap (Research Electronic Data Capture), a software toolset and workflow methodology for electronic collection and management of clinical and research data, to collect and store data. The Karolinska Institute Information Technology (KI-IT) Department will be used as a central location for data processing and management. REDCap is hosted by KI-IT in the Biomedicum (Solnavägen 9, Solna, Sweden 17165)

Data Analysis

Data analysis will be performed by the PI, co-investigators and/or key research personnel.

Quality Control and Quality Assurance

Key research personnel will be responsible for ensuring all data collected adheres to the protocol.

Data and Safety Monitoring

This study is minimal risk and all efforts will be made to ensure there are no confidentiality breaches as well as no loss of privacy.

Statistical Considerations

Power analysis This study is being conducted among several sites and thus pooled analysis will be performed. Based on the framework developed a two-sided alpha of 0.05, 250 men in each ethnicity gives 80% power to detect 10 percentage points differences in sensitivity and/or specificity of the Stockholm3 test across different ethnicities. Pooled data from several sites will allow for comparison between non-Hispanic White, Africa/Black, Asian, and Hispanic White men. Within each ethnicity group of 250 men, the same sample size gives a 90% power for detecting differences in area under curve (AUC) between Stockholm3 and PSA for detection of PC that are at least 10 percentage points (primary aim).

Goal accruement is 500 men within each race/ethnicity, interim analysis will be performed when 250 men in each race/ethnicity is enrolled.

Data Analysis Descriptive univariate statistics will be used to compare groups. Binary endpoints will be assessed with a logistic regression model. Statistical analysis will involve logistic regression modeling, AUC calculation, calibration analyses and calculation of basic performance characteristics (sensitivity, specificity and predictive values).

Regulatory Requirements

Informed Consent The participants indicate their consent to participate in the study by signing informed consents for accessing medical records, conducting genetic research and undergoing venipuncture for blood samples.

Subject Confidentiality Data used for this study will be stored in REDCaps and all data transferred between institutions will remain deidentified throughout the study.

Unanticipated Problems Any unanticipated problems will be immediately reported to the Site-specific ethical review board by designated research personnel.

ELIGIBILITY:
Inclusion Criteria:

* All men (age 45.0 - 75.0 years), regardless of race, presenting to a practicing urologist with symptoms that would lead to an evaluation for prostate cancer and who are scheduled to receive a needle biopsy of the prostate
* No prior diagnosis of prostate cancer

Exclusion Criteria:

* Men who in the three (3) months prior to study participation received any invasive urologic procedure such as biopsy, thermotherapy, microwave therapy, laser therapy, transurethral resection of the prostate (TURP), urethral catheterization, and lower genitourinary tract endoscopy (cystoscopy)
* Men who were subjected to DRE or prostate manipulation within five (5) days (120 hours) prior to blood sampling

Ages: 45 Years to 75 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologic XY sex
Study Population: The subjects will be consented for prostate biopsy as part of standard of care. No additional advertising will be used for enrollment. Patients will be identified in clinic which meet the above inclusion criteria for prostate biopsy as part of routine practice. Enrollment will start from date of IRB approval and continue until study enrollment goal. Study enrollment goal will be 2,000 men who have a self-described race/ethnicity of: African/Black (n=500), Asian (n=500), Hispanic White/Caucasian (n=500), and Non-Hispanic White/Caucasian (n=500) men.
Sampling Method: Probability Sample
Enrollment: 2152 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Gleason Grade Group 2 Prostate Cancer | On prostate biopsy immediately following PSA
  International Society of Urological Pathology Gleason Grade Group 2 Prostate Cancer. Gleason Grade Group scale is used to grade prostate cancer if found on a scale from 1 to 5. A higher score means a worse outcome.

SECONDARY OUTCOMES:
National Comprehensive Cancer Network (NCCN) unfavorable intermediate risk prostate cancer or higher risk | On prostate biopsy immediately following PSA
  National Comprehensive Cancer Network Unfavorable intermediate risk prostate cancer or higher risk. National Comprehensive Cancer Network risk stratification scores range from very low risk, low risk, intermediate risk, high risk and very high risk. Intermediate risk is stratified into favorable intermediate risk and unfavorable intermediate risk. The higher the risk the worse the outcome

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Grönberg, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (14):
- United States (13):
  - Los Angeles County, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Northwestern Medicine, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Cook County Health System, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Uropartners, Westchester, Illinois
  - Montefiore Medical Center, The Bronx, New York
  - Urology Clinics of North Texas, Dallas, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kasivisvanathan V, Rannikko AS, Borghi M, Panebianco V, Mynderse LA, Vaarala MH, Briganti A, Budaus L, Hellawell G, Hindley RG, Roobol MJ, Eggener S, Ghei M, Villers A, Bladou F, Villeirs GM, Virdi J, Boxler S, Robert G, Singh PB, Venderink W, Hadaschik BA, Ruffion A, Hu JC, Margolis D, Crouzet S, Klotz L, Taneja SS, Pinto P, Gill I, Allen C, Giganti F, Freeman A, Morris S, Punwani S, Williams NR, Brew-Graves C, Deeks J, Takwoingi Y, Emberton M, Moore CM; PRECISION Study Group Collaborators. MRI-Targeted or Standard Biopsy for Prostate-Cancer Diagnosis. N Engl J Med. 2018 May 10;378(19):1767-1777. doi: 10.1056/NEJMoa1801993. Epub 2018 Mar 18. PMID 29552975
- [Background] Gronberg H, Adolfsson J, Aly M, Nordstrom T, Wiklund P, Brandberg Y, Thompson J, Wiklund F, Lindberg J, Clements M, Egevad L, Eklund M. Prostate cancer screening in men aged 50-69 years (STHLM3): a prospective population-based diagnostic study. Lancet Oncol. 2015 Dec;16(16):1667-76. doi: 10.1016/S1470-2045(15)00361-7. Epub 2015 Nov 10. PMID 26563502
- [Background] Strom P, Nordstrom T, Aly M, Egevad L, Gronberg H, Eklund M. The Stockholm-3 Model for Prostate Cancer Detection: Algorithm Update, Biomarker Contribution, and Reflex Test Potential. Eur Urol. 2018 Aug;74(2):204-210. doi: 10.1016/j.eururo.2017.12.028. Epub 2018 Jan 10. PMID 29331214
- [Background] Moller A, Olsson H, Gronberg H, Eklund M, Aly M, Nordstrom T. The Stockholm3 blood-test predicts clinically-significant cancer on biopsy: independent validation in a multi-center community cohort. Prostate Cancer Prostatic Dis. 2019 Mar;22(1):137-142. doi: 10.1038/s41391-018-0082-5. Epub 2018 Aug 31. PMID 30171228
- [Background] Vigneswaran HT, Discacciati A, Gann PH, Gronberg H, Eklund M, Abern MR. Ethnic variation in prostate cancer detection: a feasibility study for use of the Stockholm3 test in a multiethnic U.S. cohort. Prostate Cancer Prostatic Dis. 2021 Mar;24(1):120-127. doi: 10.1038/s41391-020-0250-2. Epub 2020 Jul 8. PMID 32641739
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Potts JM, Lutz M, Walker E, Modlin C, Klein E. Trends in PSA, age and prostate cancer detection among black and white men from 1990-2006 at a tertiary care center. Cancer. 2010 Aug 15;116(16):3910-5. doi: 10.1002/cncr.25124. PMID 20564087
- [Background] Moyer VA; U.S. Preventive Services Task Force. Screening for prostate cancer: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2012 Jul 17;157(2):120-34. doi: 10.7326/0003-4819-157-2-201207170-00459. PMID 22801674
- [Background] Parekh DJ, Punnen S, Sjoberg DD, Asroff SW, Bailen JL, Cochran JS, Concepcion R, David RD, Deck KB, Dumbadze I, Gambla M, Grable MS, Henderson RJ, Karsh L, Krisch EB, Langford TD, Lin DW, McGee SM, Munoz JJ, Pieczonka CM, Rieger-Christ K, Saltzstein DR, Scott JW, Shore ND, Sieber PR, Waldmann TM, Wolk FN, Zappala SM. A multi-institutional prospective trial in the USA confirms that the 4Kscore accurately identifies men with high-grade prostate cancer. Eur Urol. 2015 Sep;68(3):464-70. doi: 10.1016/j.eururo.2014.10.021. Epub 2014 Oct 27. PMID 25454615
- [Background] de la Calle C, Patil D, Wei JT, Scherr DS, Sokoll L, Chan DW, Siddiqui J, Mosquera JM, Rubin MA, Sanda MG. Multicenter Evaluation of the Prostate Health Index to Detect Aggressive Prostate Cancer in Biopsy Naive Men. J Urol. 2015 Jul;194(1):65-72. doi: 10.1016/j.juro.2015.01.091. Epub 2015 Jan 28. PMID 25636659
- [Background] Roobol MJ, Verbeek JFM, van der Kwast T, Kummerlin IP, Kweldam CF, van Leenders GJLH. Improving the Rotterdam European Randomized Study of Screening for Prostate Cancer Risk Calculator for Initial Prostate Biopsy by Incorporating the 2014 International Society of Urological Pathology Gleason Grading and Cribriform growth. Eur Urol. 2017 Jul;72(1):45-51. doi: 10.1016/j.eururo.2017.01.033. Epub 2017 Feb 2. PMID 28162815
- [Background] Ankerst DP, Straubinger J, Selig K, Guerrios L, De Hoedt A, Hernandez J, Liss MA, Leach RJ, Freedland SJ, Kattan MW, Nam R, Haese A, Montorsi F, Boorjian SA, Cooperberg MR, Poyet C, Vertosick E, Vickers AJ. A Contemporary Prostate Biopsy Risk Calculator Based on Multiple Heterogeneous Cohorts. Eur Urol. 2018 Aug;74(2):197-203. doi: 10.1016/j.eururo.2018.05.003. Epub 2018 May 16. PMID 29778349
- [Background] Ankerst DP, Hoefler J, Bock S, Goodman PJ, Vickers A, Hernandez J, Sokoll LJ, Sanda MG, Wei JT, Leach RJ, Thompson IM. Prostate Cancer Prevention Trial risk calculator 2.0 for the prediction of low- vs high-grade prostate cancer. Urology. 2014 Jun;83(6):1362-7. doi: 10.1016/j.urology.2014.02.035. PMID 24862395
- [Background] Lichtenstein P, Holm NV, Verkasalo PK, Iliadou A, Kaprio J, Koskenvuo M, Pukkala E, Skytthe A, Hemminki K. Environmental and heritable factors in the causation of cancer--analyses of cohorts of twins from Sweden, Denmark, and Finland. N Engl J Med. 2000 Jul 13;343(2):78-85. doi: 10.1056/NEJM200007133430201. PMID 10891514
- [Background] Gronberg H, Eklund M, Picker W, Aly M, Jaderling F, Adolfsson J, Landquist M, Haug ES, Strom P, Carlsson S, Nordstrom T. Prostate Cancer Diagnostics Using a Combination of the Stockholm3 Blood Test and Multiparametric Magnetic Resonance Imaging. Eur Urol. 2018 Dec;74(6):722-728. doi: 10.1016/j.eururo.2018.06.022. Epub 2018 Jul 9. PMID 30001824
- [Background] Carroll PH, Mohler JL. NCCN Guidelines Updates: Prostate Cancer and Prostate Cancer Early Detection. J Natl Compr Canc Netw. 2018 May;16(5S):620-623. doi: 10.6004/jnccn.2018.0036. PMID 29784740
- [Background] Pepe MS, Alonzo TA. Comparing disease screening tests when true disease status is ascertained only for screen positives. Biostatistics. 2001 Sep;2(3):249-60. doi: 10.1093/biostatistics/2.3.249. PMID 12933537
- [Derived] Vigneswaran HT, Eklund M, Discacciati A, Nordstrom T, Hubbard RA, Perlis N, Abern MR, Moreira DM, Eggener S, Yonover P, Chow AK, Watts K, Liss MA, Thoreson GR, Abreu AL, Sonn GA, Palsdottir T, Plym A, Wiklund F, Gronberg H, Murphy AB; SEPTA STHLM3 Study Group. Stockholm3 in a Multiethnic Cohort for Prostate Cancer Detection (SEPTA): A Prospective Multicentered Trial. J Clin Oncol. 2024 Nov 10;42(32):3806-3816. doi: 10.1200/JCO.24.00152. Epub 2024 Jul 22. PMID 39038251